CLINICAL TRIAL: NCT03814343
Title: Comparison of Effectiveness of Topical Amphotericin B in 30% Dimethylsulphoxide and 30% Dimethylsulphoxide in Treating of Non-dermatophytes Onychomycosis: Randomized Double Blind Controlled Trial Pilot Study
Brief Title: Topical Amphotericin B in 30% Dimethylsulphoxide in Treating of Non-dermatophytes Onychomycosis
Acronym: amphotericin
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 799/2018
Record Dates: First submitted 2019-01-16; First posted 2019-01-24 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Fungal Infection; Onychomycosis; Fungus, Nail
Keywords: fungal infection; onychomycosis; amphotericin B; Dimethylsulphoxide; non-dermatophyte; randomized double blind controlled trial
MeSH Terms: conditions — Mycoses; Onychomycosis | interventions — Amphotericin B; Dimethyl Sulfoxide

STUDY DESIGN:
Intervention Model Description: Randomized double blind controlled trial pilot study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blind controlled trial between participants, drug preparing team, doctors, investigators, and outcome assessors.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active comparator (Active Comparator): 10 patients with NDMs onychomycosis treated with amphotericin B in 30% DMSO.
  Interventions: Drug: amphotericin B in 30% DMSO
- control comparator (Placebo Comparator): 10 patients with NDMs onychomycosis treated with 30% DMSO.
  Interventions: Drug: 30% DMSO

INTERVENTIONS:
Drug: amphotericin B in 30% DMSO — amphotericin B in 30% DMSO was given to patients in active comparators group for continuous 12 weeks.
  Arms: Active comparator
Drug: 30% DMSO — 30% DMSO was given to patients in placebo comparators group for continuous 12 weeks.
  Arms: control comparator

SUMMARY:
The randomized control trial study aimed to evaluate effectiveness and safety of amphotericin B in 30% DMSO solution comparing with 30% DMSO solution in NDMs onychomycosis treatment.

DETAILED DESCRIPTION:
Introduction Onychomycosis caused by non-dermatophyte molds (NDMs) have become more common in clinical practice, particularly in tropical and subtropical area. With worldwide prevalence as high as 10-24% for nail infection, more recent studies have focused on the treatment regimens for NDMs onychomycosis, especially of Neoscytalidium spp and Fusarium spp. etiology. However, there has been no consensus to-date regarding standard treatment of choice for NDMs onychomycosis.

NDMs onychomycosis was considered to be recalcitrant infection. Previous in vitro study in Malaysia reported high susceptibility of Neoscytalidium dimidiatum in amphotericin B, voriconazole, and miconazole treatment.Different therapeutic approaches such as oral antifungal agents, keratolytic agents, combined oral antifungal agents with keratolytic agents, or surgical nail avulsion, have been implemented but none has been considered a gold standard protocol in NDMs onychomycosis.

Amphotericin B is the polyene class of antimicrobial compounds. Its properties are fungicidal and have a broad spectrum with a low rate of resistance. In in vitro study, amphotericin B was reported to have better efficacy of treating N. dimidiatum infection followed by terbinafine and voricanazole. The mechanism of action is the interaction with ergosterol of fungi membrane resulting in forming permeable channels in cellular membrane of targeted fungi. This causes impairing membrane barrier function. In addition, it also causes growth inhibition. Amphotericin B is often used in treating disseminated fungal infection and visceral leishmaniasis. However, Amphotericin B can cause several side effects including nephrotocixicity, fever, chills, nausea, vomiting, headache, anemia, electrolytes imbalance (hypokalemia and hypomagnesaemia). Oral amphotercin B has poor bioavailability. Topical forms are not commonly used due to its highly lipophilic property. As a consequence, topical amphotericin B is not well absorbed through mucosa or skin resulting in low efficacy. High dose of topical amphotericin B had been developed but the results didn't work well because it caused severe adverse events such as blistering, itching, redness, peeling or severe irritation of the skin and did not even achieve the goal of treatment.

Dimethylsulphoxide (DMSO) is a promising vehicle to enhance the penetration of the drugs to animal or human skin. In addition, DMSO also has fungicidal activity. In vitro release study of amphotericin B from amphotericin B in 30% DMSO solution conducted in Siriraj Hospital revealed adequate amphotericin B concentration in the nails.

Since skin and nail infections caused by NDMs especially N. dimidiatum has been diagnosed in many countries with the majority cases being reported from Thailand, it could be implied that N. dimidiatum was endemic pathogens in this area. Published data on treatment regimens of NDMs nail infection using amphotericin B are still limited. According to the high antifungal property and low rate of drug resistance of amphotericin B, this randomized control trial study aimed to evaluate effectiveness and safety of amphotericin B in 30% DMSO solution comparing with 30% DMSO solution.

Objectives

1. To evaluate effectiveness including mycological cure of amphotericin B in 30% DMSO solution comparing with 30% DMSO solution in NDMs onychomycosis treatment
2. To evaluate safety of amphotericin B in 30% DMSO solution comparing with 30% DMSO solution in NDMs onychomycosis treatment

Material and Methods Patients Since there was no previous study that compared amphotericin B in 30% DMSO with pure 30% DMSO in treating of NDMs onychomycosis, this study designated a total of 20 patients into two groups as 10 patients with NDMs onychomycosis treated with 30% DMSO (control group) and another 10 Patients with NDMs onychomycosis treated with amphotericin B in 30% DMSO. NDMs onychomycosis was diagnosed with diagnostic criteria for NDM onychomycosis proposed by Gupta et al. Patients with any systemic or topical antifungal agents at least 3 months prior to the study were excluded from this study.

Design of medication Drugs were prepared in two solutions. First, amphotericin B (Alpharma, Denmark) was mixed with 30% DMSO (Sigma- Aldrich, Buchs, Switzerland) in 50:50 ratio. A final concentration of amphotericin B was 2 mg/ml. Later solution was pure 30% DMSO without amphotericin B. Those two final solutions had the same appearance, odor and texture. The solution will be kept in amber glass bottles with aluminum foil together with dropper. The drug regimen is to apply 1-3 drops of the solution once a day to each affected nail and briefly let the solution evaporate before continuing their usual activities.

Treatment, Follow-up and measurement A randomized control trial study conducted in outpatient nail clinic, Siriraj Hospital. Patients will be divided into two groups by mixed block of randomization. First groups will be treated with amphotericin B in 30% DMSO solution. Another group will be given only 30% DMSO solution. Each patient is subjected to continuously apply his/ her own drugs followed instruction given for 12 weeks. They will be followed up at 12 weeks, 24 weeks and 36 weeks for re-evaluation of clinical, mycological laboratories, adherence to the drug and adverse events. Effectiveness was evaluated by clinical improvement and mycological cure as well as median time to mycological cure. Clinical evaluation would be assessed by two treatment-blind dermatologists. Regarding mycological cure, it was defined as negative KOH and fungal culture. Data were analyzed using PASW Statistics version 18 (SPSS, Inc., Chicago, IL, USA).

Duration of study: 1 year

Study design: Randomized double blind control trial

ELIGIBILITY:
Inclusion Criteria:

1. Patients with non-dermatophyte onychomycosis.
2. Patients aged more than 18 years.
3. Patients has not been treated with any oral/ IV/ topical antifungal therapy within 36 weeks before enrolled.

Exclusion Criteria:

1. Patients had concomitant nail diseases.
2. Immunocompromised host.
3. Patients with dermatophyte onychomycosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2020-11-15 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
Effectiveness of amphotericin B in 30% DMSO solution comparing with 30% DMSO solution in NDMs onychomycosis treatment | 36 weeks
  Effectiveness was evaluated by patients who had negative on mycological laboratory (mycological cure) as percentage.
Median time to mycological cure of patients with amphotericin B in 30% DMSO solution comparing with 30% DMSO solution in NDMs onychomycosis treatment | 36 weeks
  Median time to mycological cure were defined as time (days, months or years) that had negative on mycological laboratory

SECONDARY OUTCOMES:
Clinical cure of amphotericin B in 30% DMSO solution comparing with 30% DMSO solution in NDMs onychomycosis treatment | 36 weeks
  Clinical cure was defined as the patients had complete clinical improvement or having <10% nail involvement.
Median time to clinical cure of patients with amphotericin B in 30% DMSO solution comparing with 30% DMSO solution in NDMs onychomycosis treatment | 36 weeks
  Median time to clinical cure were defined as time (days, months or years) that had clinical improvement of the affected nails.
Evaluate side effects of amphotericin B in 30% DMSO solution comparing with 30% DMSO solution in NDMs onychomycosis treatment | 12 weeks
  Side effects was assessed by the percentage of patients developed any side effect such as erythema, burning sensation, pain.

CONTACTS AND LOCATIONS:
Overall Officials: Sumanas Bunyaratavej, MD, Principal Investigator — Mahidol University; Charussri Leeyaphan, MD, Study Director — Mahidol University
Locations (1):
- Department of Dermatology Siriraj Hospital, Bangkoknoi, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Butani D, Yewale C, Misra A. Amphotericin B topical microemulsion: formulation, characterization and evaluation. Colloids Surf B Biointerfaces. 2014 Apr 1;116:351-8. doi: 10.1016/j.colsurfb.2014.01.014. Epub 2014 Jan 19. PMID 24521698
- [Result] Downs AM, Lear JT, Archer CB. Scytalidium hyalinum onychomycosis successfully treated with 5% amorolfine nail lacquer. Br J Dermatol. 1999 Mar;140(3):555. doi: 10.1046/j.1365-2133.1999.02739.x. No abstract available. PMID 10233295
- [Result] Cursi IB, Silva RT, Succi IB, Bernardes-Engemann AR, Orofino-Costa R. Onychomycosis due to Neoscytalidium treated with oral terbinafine, ciclopirox nail lacquer and nail abrasion: a pilot study of 25 patients. Mycopathologia. 2013 Feb;175(1-2):75-82. doi: 10.1007/s11046-012-9580-5. Epub 2012 Sep 14. PMID 22976905
- [Result] Tosti A, Piraccini BM, Lorenzi S. Onychomycosis caused by nondermatophytic molds: clinical features and response to treatment of 59 cases. J Am Acad Dermatol. 2000 Feb;42(2 Pt 1):217-24. doi: 10.1016/S0190-9622(00)90129-4. PMID 10642676
- [Result] Welsh O, Vera-Cabrera L, Welsh E. Onychomycosis. Clin Dermatol. 2010 Mar 4;28(2):151-9. doi: 10.1016/j.clindermatol.2009.12.006. PMID 20347657
- [Result] Gupta AK, Drummond-Main C, Cooper EA, Brintnell W, Piraccini BM, Tosti A. Systematic review of nondermatophyte mold onychomycosis: diagnosis, clinical types, epidemiology, and treatment. J Am Acad Dermatol. 2012 Mar;66(3):494-502. doi: 10.1016/j.jaad.2011.02.038. Epub 2011 Aug 4. PMID 21820203
- [Result] Bunyaratavej S, Prasertworonun N, Leeyaphan C, Chaiwanon O, Muanprasat C, Matthapan L. Distinct characteristics of Scytalidium dimidiatum and non-dermatophyte onychomycosis as compared with dermatophyte onychomycosis. J Dermatol. 2015 Mar;42(3):258-62. doi: 10.1111/1346-8138.12768. Epub 2015 Jan 13. PMID 25639524
- [Result] Bunyaratavej S, Leeyaphan C, Rujitharanawong C, Surawan TM, Muanprasat C, Matthapan L. Efficacy of 5% amorolfine nail lacquer in Neoscytalidium dimidiatum onychomycosis. J Dermatolog Treat. 2016 Aug;27(4):359-63. doi: 10.3109/09546634.2015.1109029. Epub 2015 Nov 11. PMID 26471716
- [Result] Gupta AK, Paquet M, Simpson FC. Therapies for the treatment of onychomycosis. Clin Dermatol. 2013 Sep-Oct;31(5):544-54. doi: 10.1016/j.clindermatol.2013.06.011. PMID 24079583
- [Result] Machouart M, Menir P, Helenon R, Quist D, Desbois N. Scytalidium and scytalidiosis: what's new in 2012? J Mycol Med. 2013 Mar;23(1):40-6. doi: 10.1016/j.mycmed.2013.01.002. Epub 2013 Feb 15. PMID 23416171
- [Result] James JE, Santhanam J, Lee MC, Wong CX, Sabaratnam P, Yusoff H, Tzar MN, Razak MF. In Vitro Antifungal Susceptibility of Neoscytalidium dimidiatum Clinical Isolates from Malaysia. Mycopathologia. 2017 Apr;182(3-4):305-313. doi: 10.1007/s11046-016-0085-5. Epub 2016 Nov 4. PMID 27815659
- [Result] Lurati M, Baudraz-Rosselet F, Vernez M, Spring P, Bontems O, Fratti M, Monod M. Efficacious treatment of non-dermatophyte mould onychomycosis with topical amphotericin B. Dermatology. 2011;223(4):289-92. doi: 10.1159/000335093. Epub 2012 Jan 10. PMID 22236569
- [Result] Hussain A, Samad A, Singh SK, Ahsan MN, Haque MW, Faruk A, Ahmed FJ. Nanoemulsion gel-based topical delivery of an antifungal drug: in vitro activity and in vivo evaluation. Drug Deliv. 2016;23(2):642-47. doi: 10.3109/10717544.2014.933284. Epub 2014 Jul 11. PMID 25013957
- [Result] Zaioncz S, Khalil NM, Mainardes RM. Exploring the Role of Nanoparticles in Amphotericin B Delivery. Curr Pharm Des. 2017;23(3):509-521. doi: 10.2174/1381612822666161027103640. PMID 27799043
- [Result] Ungpakorn R, Lohaprathan S, Reangchainam S. Prevalence of foot diseases in outpatients attending the Institute of Dermatology, Bangkok, Thailand. Clin Exp Dermatol. 2004 Jan;29(1):87-90. doi: 10.1111/j.1365-2230.2004.01446.x. PMID 14723731